CLINICAL TRIAL: NCT03604419
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Dose Cohort Study to Evaluate the Efficacy and Safety of Twelve Once-weekly Subcutaneous Doses of PB-119 to Patients With Type 2 Diabetes Mellitus (T2DM) Not Well-controlled by Metformin Monotherapy
Brief Title: Dose-finding of PB-119 Administered Subcutaneously Once Weekly Versus Placebo in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PegBio Co., Ltd. (Other)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PB119202
Record Dates: First submitted 2018-05-25; First posted 2018-07-27 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PB-119 100 μg (Experimental): PB-119 100 μg subcutaneous (SC) once weekly (QW) + Metformin oral (p.o.) Glucophage® (stable dosage)
  Interventions: Drug: PB-119 150 μg+ Glucophage®; Drug: PB-119 200 μg+ Glucophage®; Drug: PB-119 placebo + Glucophage®
- PB-119 150 μg (Experimental): PB-119 150 μg SC QW + Metformin oral (p.o.) Glucophage® (stable dosage)
  Interventions: Drug: PB-119 100 μg+ Glucophage®; Drug: PB-119 200 μg+ Glucophage®; Drug: PB-119 placebo + Glucophage®
- PB-119 200 μg (Experimental): PB-119 200 μg SC QW + Metformin oral (p.o.) Glucophage® (stable dosage)
  Interventions: Drug: PB-119 100 μg+ Glucophage®; Drug: PB-119 150 μg+ Glucophage®; Drug: PB-119 placebo + Glucophage®
- PB-119 Placebo (Placebo Comparator): PB-119 Placebo SC QW + Metformin oral (p.o.) Glucophage® (stable dosage)
  Interventions: Drug: PB-119 100 μg+ Glucophage®; Drug: PB-119 150 μg+ Glucophage®; Drug: PB-119 200 μg+ Glucophage®

INTERVENTIONS:
Drug: PB-119 100 μg+ Glucophage® — Each patient will subsequently be randomized within the designated cohort to active drug or placebo
  Arms: PB-119 150 μg; PB-119 200 μg; PB-119 Placebo
Drug: PB-119 150 μg+ Glucophage® — Each patient will subsequently be randomized within the designated cohort to active drug or placebo
  Arms: PB-119 100 μg; PB-119 200 μg; PB-119 Placebo
Drug: PB-119 200 μg+ Glucophage® — Each patient will subsequently be randomized within the designated cohort to active drug or placebo
  Arms: PB-119 100 μg; PB-119 150 μg; PB-119 Placebo
Drug: PB-119 placebo + Glucophage® — Each patient will subsequently be randomized within the designated cohort to active drug or placebo
  Arms: PB-119 100 μg; PB-119 150 μg; PB-119 200 μg

SUMMARY:
A phase 2, multicenter study to evaluate the efficacy and safety of twelve once weekly subcutaneous doses of PB-119 to patients with type 2 diabetes mellitus (T2DM) not well-controlled by metformin mono therapy.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel dose cohort, multiple dose study to evaluate the efficacy, safety, and tolerability of different doses of PB-119 to patients with T2DM not well-controlled by metformin monotherapy. Patients will be assessed for eligibility over a 2 week screening period prior to a 4-week run-in period and a 12-week double-blind treatment period.A phase 2, multicenter, randomized, double-blind, placebo-controlled, parallel dose cohort study to evaluate the efficacy and safety of twelve once weekly subcutaneous doses of PB-119 to patients with type 2 diabetes mellitus (T2DM) not well-controlled by metformin monotherapy The eligible patients will be randomized to 1 of 3 dose cohorts (A, B, or C). Each patient will subsequently be randomized within the designated cohort to 1) active drug or placebo at a 3:1 active drug:placebo ratio and 2) exclusion from or inclusion in the pharmacokinetic (PK) blood sample collection subgroup at a 3:1 excluded:included ratio

ELIGIBILITY:
Inclusion Criteria:

1. Patients in whom T2DM has been diagnosed according to 2018 American Diabetes Association T2DM diagnostic criteria, have made lifestyle modifications (ie, diet and exercise) for at least 3 months prior to Screening, and have been taking metformin for at least 3 months before Screening with a stable dosage for at least 8 weeks (stable dosage is defined as metformin dosage ≥1500 mg/day or maximum tolerated dose).
2. Males and/or females between the ages of ≥18 and ≤70 years at Screening
3. HbA1c ≥7.5% and ≤11% at Screening and at Week -1, Visit 3.1;
4. FPG ≥126 and ≤240 mg/dL (≥7.0 and ≤13.3 mmol/L) at Screening and at Week -1, Visit 3.1;
5. Body mass index (BMI) ≥18.5 and ≤40.0 kg/m2 at Screening, with inclusion of patients with BMIs at the lower end of the range enrolled into the study to enable comparisons across BMI range;

Exclusion Criteria:

1. Medical history or current diagnosis of:

   1. Type 1 diabetes mellitus, diabetes caused by pancreas injury or by other diseases (like acromegaly or Cushing syndrome);
   2. Diabetes acute complication, like ketoacidosis or hyperosmolar coma;
   3. Diagnosed proliferative retinopathy;
   4. 3 instances of severe hypoglycemia (events during which the patient required the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions; episodes may be associated with sufficient neuroglycopenia to have induced seizure or coma) in the 6 months prior to Screening;
   5. Significant vascular disease;
2. Current/ongoing diagnosis of any type of malignant tumor or evidence of recurrence in the 6 months prior to Screening (patients who have been stable for ≥6 months or those who have had basal or squamous cell skin cancers removed and have no evidence of recurrence will not be excluded). Patients with a medical history of any other type of cancer in the last 5 years prior to Screening will be excluded;
3. Severe cardiovascular diseases occurring within 6 months prior to Screening (eg, congestive heart disease, myocardial infarction, acute coronary syndrome, apoplexy, transient ischemic attack);

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-07-23 (Actual)

PRIMARY OUTCOMES:
The change from baseline value of HbA1c will be compared between treatments | From Baseline to end of treatment (up to Week 12)

SECONDARY OUTCOMES:
The change from baseline value of Fasting Plasma Glucose at Weeks 2, 4, 8, and 12 | From Baseline to end of treatment (up to Week 12)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Pharmacology of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park EJ, Choi J, Lee KC, Na DH. Emerging PEGylated non-biologic drugs. Expert Opin Emerg Drugs. 2019 Jun;24(2):107-119. doi: 10.1080/14728214.2019.1604684. Epub 2019 Apr 19. PMID 30957581